CLINICAL TRIAL: NCT04547413
Title: Prospective Cohort Trial To Assess Acceptability and Efficacy of an Adapted STI/HIV Intervention Behavioral Intervention Program in a Population of US Army Personnel and Their Medical Beneficiaries - Execution Phase
Brief Title: STI/HIV Intervention Behavioral Intervention Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Madigan Army Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RV567
Record Dates: First submitted 2020-08-21; First posted 2020-09-14 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Sexually Transmitted Infections
Keywords: STI; HIV; syphilis; gonorrhea; chlamydia; mycoplasma genitalium
MeSH Terms: conditions — Sexually Transmitted Diseases; Syphilis; Gonorrhea; Chlamydia Infections | interventions — Mass Screening

STUDY DESIGN:
Intervention Model Description: This is a randomized, controlled trial of a behavioral intervention designed to increase the use of safer sexual practices and to reduce incident STi rates. The intervention is a 2-hour class based program and therefore is not blinded. Outcome measures of sexual behavior and incident STIs will be measured at 6 and 12 months after the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm (No Intervention): Control Arm will will complete a total of three visits:
  Visit 1 (Day 1): Recruitment/Baseline Biological Testing, if needed; completion of baseline study surveys including Knowledge Assessment
  Monthly: Prevention Maintenance Intervention Messages from months 2-11
  Visit 3 (Day 180): 6 Month Follow-up biological testing and study survey
  Visit 4 (Day 365): 12 Month Follow-up biological testing and study surveys
- Intervention Arm (Active Comparator): Intervention Arm will will complete a total of four visits:
  Visit 1 (Day 1): Recruitment/Baseline Biological Testing, if needed; completion of baseline study surveys including Knowledge Assessment
  Visit 2 (Day 2-30): Group Intervention Session, Feedback form, and post-intervention knowledge assessment (for intervention arm only)
  Monthly: Prevention Maintenance Intervention Messages from months 2-11
  Visit 3 (Day 180): 6 Month Follow-up biological testing and study survey
  Visit 4 (Day 365): 12 Month Follow-up biological testing and study surveys
  Interventions: Behavioral: STI/HIV Intervention Behavioral Intervention Program

INTERVENTIONS:
Behavioral: STI/HIV Intervention Behavioral Intervention Program — In addition to standard of care STi/HIV counselling, participants in the intervention arm will also attend a 2-hour educational class and will receive monthly SMS/text messages to reinforce the content of the class.
  Other Names: KISS (Knocking out Infections through Safer sex and Screening
  Arms: Intervention Arm

SUMMARY:
The hypothesis is that a behavioral intervention tool adapted for the US military population will be acceptable and associated with a decrease in incident sexually transmitted infection (STI)/HIV rates and high-risk sexual behaviors, and increased self-reported condom use compared to the standard of care at the Joint Base Lewis-McChord (JBLM) Preventive Medicine clinic and the Fort Bragg Department of Public Health (part of Womack Army Medical Center).

DETAILED DESCRIPTION:
This is the Execution Phase which will be conducted as a multi-site randomized controlled trial. A previous Formative Phase study was conducted under a separate protocol which has been completed with preliminary data indicating positive outcomes. Participants in both arms will meet the same inclusion/exclusion criteria and will be randomized into the intervention and control arms at a ratio of 1:1.

The intervention arm will receive the KISS (Knocking out Infections through Safer sex and Screening) intervention program in addition to standard STI prevention counselling routinely provided by military medical treatment facilities. The control arm will receive only standard STI prevention counselling. Both arms will receive follow-up educational messages via short message service (SMS)/text messaging monthly for 10 months, and have follow-up study visits at 6 months and 12 months.

The KISS intervention is a 2-hour, small group (6-12 individuals) class-based interactive, educational session based on Social Cognitive Theory and the Theory of Gender and Power. The intervention is an adaptation of the HORIZONS intervention, which has shown efficacy are reducing sexual risk behavior and incident STIs among adolescents in the USA. HORIZONS has been reviewed by the U.S. Centers for Disease Control (CDC) Prevention Synthesis Research team and designated a CDC top-tier (Tier I) evidence-based intervention (EBI).

To enroll in the study, participants must be categorized as "high risk" as determined by a positive test for an STI within the previous 180 days or has had STI screening during this time frame (specifically gonorrhea (GC), chlamydia (CT), M. genitalium, syphilis and/or HIV).

Study subjects will be recruited from Madigan Army Medical Center (Madigan) Preventive Medicine Clinic and the Womack Army Medical Center (Womack) Preventive Medicine Clinic in Ft. Bragg, North Carolina (NC). In addition, promotional flyers for recruitment will be placed in public areas on both bases, and will be promoted through approved social media channels. Subjects may also refer up to 5 friends or colleagues for screening.

Participants enrolled in the intervention arm will complete a total of four visits and those in the control arm will complete a total of three visits. Over the course of the study, participants in both groups will be asked to provide biological specimens and complete knowledge/behavioral surveys three times (at baseline, 6 and at 12 months). Those in the intervention group will also attend the KISS EBI (Evidence Based Intervention) program. Both arms will receive monthly (months 2-11) follow up text messages, but the content will defer between the two arms. Those in the intervention arm, will receive SMS/text messages targeting prevention maintenance interventions (PMI) messages reiterating information received during the EBI session. Those in the control arm, will receive SMS/text messages that will contain general health information.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 - 30 years
2. Army active duty or Army medical beneficiary
3. Eligible to receive care at a military healthcare clinic for at least 12 months from enrollment
4. HIV negative
5. Not scheduled for military deployment or transfer within 3 months of enrolment
6. Not pregnant, regardless of marital status
7. Not trying to become pregnant or impregnate a partner, regardless of marital status
8. Be classified as "high risk" either through a positive STI diagnosis in the last 180 days or has had STI screening during this timeframe.
9. Self reports vaginal, oral, and/or anal sexual contact in the last 30 days.

Exclusion Criteria:

1. Under 18 or over 30 years of age
2. Not Army active duty or Army medical beneficiary
3. Not eligible to receive care at a military healthcare clinic for study duration (next 12 months)
4. HIV positive
5. Military deployment or transfer scheduled within 3 months of enrollment
6. Are pregnant, regardless of marital status
7. Are trying to become pregnant or impregnate someone, regardless of marital status
8. Has not had a positive STI diagnosis or STI screening within the last 180 days
9. Does not self-report vaginal, anal, and/or oral sexual contact in the last 30 days

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 155 (Actual)
Dates: Start 2020-11-04 (Actual); Primary Completion 2024-03-10 (Actual); Study Completion 2024-03-10 (Actual)

PRIMARY OUTCOMES:
Incident sexually transmitted infections | 12 months
  Biological testing for syphilis, chlamydia trachomatis, neisseria gonorrhea, mycoplasma genitalium, and HIV
Acceptability of the intervention | immediately after the intervention
  participant feedback and rating of the intervention session

SECONDARY OUTCOMES:
Number of sexual partners | 12 months
  self-report by questionnaire
Proportion of sexual encounters protect by condom use | 12 months
  self-report by questionnaire

OTHER OUTCOMES:
Change in Knowledge about STIs, HIV and prevention: post-intervention | Baseline and immediately after the intervention
  Completion of a 20-item standardized questionnaire on STI/HIV transmission, symptoms, and prevention methods
Change in Knowledge about STIs, HIV and prevention: retention at 6 months | Baseline, immediately after the intervention, and at 6 months
  Completion of a 20-item standardized questionnaire on STI/HIV transmission, symptoms, and prevention methods
Change in Knowledge about STIs, HIV and prevention: retention at 12 months | Baseline, immediately after the intervention, and at 12 months
  Completion of a 20-item standardized questionnaire on STI/HIV transmission, symptoms, and prevention methods

CONTACTS AND LOCATIONS:
Overall Officials: Tatjana Calvano, MD, Principal Investigator — Madigan Army Medical Center
Locations (2):
- United States (2):
  - Ft. Bragg, Fayetteville, North Carolina
  - Madigan Army Medical Center, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: No
Requests for data sharing may be considered on a case-by-case basis

REFERENCES:
- [Derived] Romo ML, Moreland SC, Yates AM, Crowell TA, Sevilla M, MacArthur JL, Faestel P, Kunz A, Ake JA, Calvano T, Colby DJ. Prevalence of Urogenital Mycoplasma genitalium Infection at 2 US Army Medical Facilities. Sex Transm Dis. 2024 May 1;51(5):367-373. doi: 10.1097/OLQ.0000000000001947. Epub 2024 Feb 10. PMID 38346403
- [Derived] Kunz A, Moodley A, Colby DJ, Soltis M, Robb-McGrath W, Fairchok A, Faestel P, Jungels A, Bender AA, Kamau E, Wingood G, DiClemente R, Scott P. Feasibility, acceptability, and short-term impact of a brief sexually transmitted infection intervention targeting U.S. Military personnel and family members. BMC Public Health. 2022 Apr 2;22(1):640. doi: 10.1186/s12889-022-13096-x. PMID 35366848